CLINICAL TRIAL: NCT03327818
Title: Obstetric Hysterectomy Versus Conservative Surgery for Management of Patients With Morbidly Adherent Placenta as Regard Maternal Morbidity and Mortality
Brief Title: Comparison Between Hysterectomy and Conservative Management in Treatment of Placenta Accreta Regarding Maternal Complication
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Wessam Sayed Mohamed, Malames Mahmoud Faisal ,MD, Ain Shams Maternity Hospital
Other Study IDs: N01MH90003 (NIH)
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conservative surgery group
  Interventions: Procedure: uterine conservative study
- hysterectomy group
  Interventions: Procedure: hysterectomy

INTERVENTIONS:
Procedure: hysterectomy
  Groups: hysterectomy group
Procedure: uterine conservative study
  Groups: conservative surgery group

SUMMARY:
AIM OF THE WORK The aim of the study is to compare the maternal morbidity and mortality between obstetric hysterectomy and conservative surgery for pregnant ladies > 28 weeks with placenta accreta during caesarean section at Ain Shams University Maternity Hospital in the last five years and prospective study in the next six months.

Hypothesis In women with placenta accrete undergoing hysterectomy may be similar to conservative surgery as regard maternal morbidity and mortality.

DETAILED DESCRIPTION:
The study included all cases of placenta accreta that were diagnosed preoperative or intra-operative and treated by conservative surgery or by hysterectomy during caesarean section between January 2011 to December 2015 at Ain Shams University Maternity Hospital and from July 2016 to January 2017.

The collected data will be categorized according to the way of management and will be analyzed regarding:

Mortality rates.

Intraoperative morbidities:

Blood loss and it's amount and need for transfusion. Amount of blood and blood products transferred. Injury to adjacent organs eg: bladder or bowel injury.

Early postoperative morbidities:

Blood and blood product transfusion Length of maternal Hospital admission post operative Acquiring intensive care unit admission and identifying the cause and duration Wound sepsis Septic shock Peritonitis DVT Acute pulmonary embolism Hysterectomy after conservative management and its indication Wound dehiscence Burst abdomen

Late postoperative morbidities:

Anemia Recurrence of placenta accretes in next pregnancy. Hysterectomy after conservative management and its indication Uterine necrosis Fistula eg. urinary fistula

ELIGIBILITY:
Inclusion Criteria:

* Women admitted for elective caesarean section. Pregnant women more than 28weeks of gestation. Women with no associated medical diseases eg. DM, PET. Pre-operatively Hemodynamically stable women. Women diagnosed with placenta accrete either preoperative or accidentally discovered intraoperative.

Exclusion Criteria:

* Pregnant women less than 28weeks of gestation. Women with associated medical co-morbidity eg bleeding tendency eg: DM, PET.

Ages: 14 Years to 55 Years | Sex: Female
Age Groups: Child, Adult
Study Population: all cases of placenta accreta present in Ain shams university maternity hospital from 2011 to 2015 and from July 2016 to January 2017
Sampling Method: Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
maternal morbidity | 24 hours post operative